CLINICAL TRIAL: NCT06284772
Title: FINRISK 2002 Re-examination
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Teemu Niiranen, Professor, University of Turku
Other Study IDs: 4457/2023
Record Dates: First submitted 2024-02-20; First posted 2024-02-29 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-02

CONDITIONS: Cardiometabolic Syndrome; Cardiovascular Diseases
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases | interventions — Surveys and Questionnaires; Nutrition Surveys

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal samples for 2500 individuals. Serum and plasma samples for 269 individuals who took part in the health examination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- FINRISK 2002 re-examination cohort: All still-living FINRISK 2002 participants (~6000) were invited do participate in a re-examination >20 years after the initial fecal sampling. 2500 took part in the study.
  Interventions: Other: Questionnaire and fecal sampling
- FINRISK 2002 re-examination health examination: The ~800 still-living participants from the Turku and Loimaa area were asked to participate in a health examination. 269 individuals took part in the health examination.
  Interventions: Other: Questionnaire and fecal sampling; Other: Health examination

INTERVENTIONS:
Other: Questionnaire and fecal sampling — The participants will be mailed a fecal collection kit and a 20-page health questionnaire. This questionnaire will include the similar questions concerning health, lifestyles, and diet as in 2002.
Other: Health examination — This examination will include measurements for anthropometrics, cognition (MoCA, Stroop, DSST), and blood pressure. The participants will undergo blood draw for laboratory analyses of CMD risk factors, such as blood lipids, glucose metabolism (fasting glucose, HbA1c, and fasting insulin), liver enzymes (GGT, ALT, and AST), inflammation (hs-CRP), and cardiac markers (proBNP and hs-TnI). We will perform ultrasound imaging for hepatic fibrosis.
  Groups: FINRISK 2002 re-examination health examination

SUMMARY:
The project aims to fill in the existing gaps in the study of the microbiome as a cardiometabolic driver 1) by determining the key demographic, environmental, genetic, dietary, and metabolic correlates of long-term within-individual microbiome and microbial metabolite changes; and 2) by assessing how the gut microbiome, microbial metabolites, and their long-term changes are prospectively related to the risk factors, surrogate markers, and overt outcomes of CMD. To achieve this goal, repeat stool samples will be collected of ~2300 Finnish individuals who gave stool samples in the year 2002. In addition, ~300 individuals will undergo a in-depth health examination in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Participation in FINRISK 2002 fecal sampling

Ages: 47 Years to 96 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The FINRISK 2002 cohort (N=7,237 participants with sequenced fecal samples) was originally examined in 2002. The FINRISK 2002 cohort is a random sample of the Finnish population, aged 25-74 years in the year 2002, from 6 geographic regions in Finland.
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Gut microbiome change between 2002-2024 | 2002-2024
  Individual-level changes in the metagenome-sequenced gut microbiome between 2002 and 2024. The microbiome indices of interest are:
  1. Alpha diversity
  2. Beta diversity
  3. Taxonomy

SECONDARY OUTCOMES:
Correlates of gut microbiome change between 2002-2024 | 2002-2024
  Questionnaire-, biochemistry-, and health examination-derived correlates of gut microbiome change between 2002-2024.

CONTACTS AND LOCATIONS:
Overall Officials: Teemu Niiranen, MD, Principal Investigator — Department of Internal Medicine, University of Turku
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borodulin K, Tolonen H, Jousilahti P, Jula A, Juolevi A, Koskinen S, Kuulasmaa K, Laatikainen T, Mannisto S, Peltonen M, Perola M, Puska P, Salomaa V, Sundvall J, Virtanen SM, Vartiainen E. Cohort Profile: The National FINRISK Study. Int J Epidemiol. 2018 Jun 1;47(3):696-696i. doi: 10.1093/ije/dyx239. No abstract available. PMID 29165699
- [Background] Salosensaari A, Laitinen V, Havulinna AS, Meric G, Cheng S, Perola M, Valsta L, Alfthan G, Inouye M, Watrous JD, Long T, Salido RA, Sanders K, Brennan C, Humphrey GC, Sanders JG, Jain M, Jousilahti P, Salomaa V, Knight R, Lahti L, Niiranen T. Taxonomic signatures of cause-specific mortality risk in human gut microbiome. Nat Commun. 2021 May 11;12(1):2671. doi: 10.1038/s41467-021-22962-y. PMID 33976176